CLINICAL TRIAL: NCT00349648
Title: Conservative or Operative Treatment for the Shoulder Impingement Syndrome? A Randomized Controlled Trial of 140 Patients Followed Up for Two Years.
Brief Title: Conservative or Operative Treatment for the Shoulder Impingement Syndrome?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kanta-Häme Central Hospital (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IMP-E9/2001-140
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2006-07-07 (Estimated); Status verified 2006-07

CONDITIONS: Shoulder Impingement Syndrome
Keywords: subacromial; impingement; acromioplasty; physiotherapy
MeSH Terms: conditions — Shoulder Impingement Syndrome

INTERVENTIONS:
Procedure: acromioplasty

SUMMARY:
Study hypothesis: The impingement syndrome of the rotator cuff is a common cause of shoulder pain for which the most effective treatment is unknown. Steroid injections and anti-inflammatory analgetics are considered as effective methods. Physiotherapy and acromioplasty are commonly used treatments.

Hypothesis: Arthroscopy and acromioplasty in addition to conservative treatment is equally effective as conservative treatment alone for shoulder impingement syndrome.

DETAILED DESCRIPTION:
The aim of this study was to examine the effectiveness of arthroscopic acromioplasty in the treatment of the shoulder impingement syndrome. Nonoperative treatment consisted of information given by a trained physiotherapist. The patients were supervised with a progressive programme to improve the mobility and muscle strength of the shoulder region which was regularly controlled. The exercises aimed at strengthening the stabilising muscles of the glenohumeral joint (m. trapezius, m. deltoides, m. supraspinatus and m. infraspinatus) and activating the decompressive muscles of the the subacromial space (m. teres major and minor, m. subscapularis). The programme lasted for three months. In addition the patients were given advice for daily home exercise.

In the surgical group the patients underwent an arthroscopic examination and acromioplasty done by one experienced orthopaedic specialist. Postoperatively the patients received similar physiotherapeutical information and training programme than in the conservative treatment group.

The follow-up evaluations were performed at 3, 6 and 12 months from the beginning of each treatment in addition at 24 months counted from the randomization. A trained research physiotherapist who was blinded to the treatment group and had not been involved in their treatment performed a standardized assessment of all patients. The range of motion, muscle strengths and Neer´s tests were recorded. At each evaluation the patients completed a structured questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* a positive clinical Neer's test
* shoulder pain resistant to rest
* shoulder pain resistant to anti-inflammatory drugs
* shoulder pain resistant to subacromial steroid injections
* shoulder pain resistant to ordinary physiotherapy with a minimum history of three months

Exclusion Criteria:

* glenohumeral or acromioclavicular arthritis
* glenohumeral instability
* total rupture of the rotator cuff
* cervical syndrome
* adhesive capsulitis
* neuropathy of the shoulder region

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140
Dates: Start 2001-03; Study Completion 2006-07

PRIMARY OUTCOMES:
shoulder pain in visual analogue scale (VAS) of 0-10 at two years after randomization

SECONDARY OUTCOMES:
pain at night
disability
ability to work
ranges of motion
cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Saara Ketola, Principal Investigator — Kanta-Häme Central Hospital
Locations (1):
- Kanta-Häme Central Hospital, Hämeenlinna, Finland

REFERENCES:
- [Background] Brox JI, Staff PH, Ljunggren AE, Brevik JI. Arthroscopic surgery compared with supervised exercises in patients with rotator cuff disease (stage II impingement syndrome). BMJ. 1993 Oct 9;307(6909):899-903. doi: 10.1136/bmj.307.6909.899. PMID 8241852
- [Background] Green S, Buchbinder R, Glazier R, Forbes A. Interventions for shoulder pain. Cochrane Database Syst Rev. 2000;(2):CD001156. doi: 10.1002/14651858.CD001156. PMID 10796418
- [Background] Haahr JP, Ostergaard S, Dalsgaard J, Norup K, Frost P, Lausen S, Holm EA, Andersen JH. Exercises versus arthroscopic decompression in patients with subacromial impingement: a randomised, controlled study in 90 cases with a one year follow up. Ann Rheum Dis. 2005 May;64(5):760-4. doi: 10.1136/ard.2004.021188. PMID 15834056
- [Background] Leroux JL, Codine P, Thomas E, Pocholle M, Mailhe D, Blotman F. Isokinetic evaluation of rotational strength in normal shoulders and shoulders with impingement syndrome. Clin Orthop Relat Res. 1994 Jul;(304):108-15. PMID 8020202
- [Background] Neer CS 2nd. Anterior acromioplasty for the chronic impingement syndrome in the shoulder: a preliminary report. J Bone Joint Surg Am. 1972 Jan;54(1):41-50. No abstract available. PMID 5054450
- [Background] Neer CS 2nd. Impingement lesions. Clin Orthop Relat Res. 1983 Mar;(173):70-7. No abstract available. PMID 6825348